CLINICAL TRIAL: NCT06772233
Title: A Phase II, Open-label, Multicenter, Randomized Controlled Clinical Trial Comparing Regorafenib Combined With Envafolimab to Physician's Choice in Patients With Metastatic Gastrointestinal Stromal Tumors Harboring KIT Exon 17 Mutations Refractory to Standard Treatment.
Brief Title: A Study of Regorafenib Combined With Envafolimab for Metastatic Gastrointestinal Stromal Tumors With Kit Gene Exon 17 Mutation That Failed Standard Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIST 006
Record Dates: First submitted 2024-12-30; First posted 2025-01-13 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Gastrointestinal Stromal Tumors (GIST)
Keywords: gastrointestinal stromal tumors, KIT exon 17 mutations
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — envafolimab; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- regorafenib combined with envafolimab (Experimental): * Regorafenib: Specification: 40 mg/tablet Dosage: 120 mg, taken orally once daily for 3 weeks, followed by 1 week off, until disease progression or intolerable toxicity occurs.
  * Envafolimab: Specification: 200 mg/vial Dosage: 200 mg, administered via subcutaneous injection once every 2 weeks, until disease progression or intolerable toxicity occurs.
  Interventions: Drug: regorafenib combined with envafolimab
- Physician's choice (Active Comparator): The governing principle for physician decision-making in the control group was selection based on prior medication tolerability, genotype, etc.:
  1. Continued maintenance therapy with the originally effective TKI at the same dose: The patient achieved at least stable disease (SD) or partial response (PR) during prior treatment, with progression-free survival (PFS) exceeding 6 months, and the adverse reactions were tolerable.
  2. Combination therapy with two TKIs: Different drugs were selected for maintenance based on distinct actionable mutations identified in the patient's tissue or peripheral blood genetic testing, OR a combination of drugs previously effective and well-tolerated was used, OR the combination therapy was chosen by referencing past tolerability.
  Interventions: Drug: Control Group

INTERVENTIONS:
Drug: regorafenib combined with envafolimab — -Regorafenib: Specification: 40 mg/tablet Dosage: 120 mg, taken orally once daily for 3 weeks, followed by 1 week off, until disease progression or intolerable toxicity occurs.
  * Envafolimab:
  Specification: 200 mg/vial Dosage: 200 mg, administered via subcutaneous injection once every 2 weeks, until disease progression or intolerable toxicity occurs.
  Arms: regorafenib combined with envafolimab
Drug: Control Group — The governing principle for physician decision-making in the control group was selection based on prior medication tolerability, genotype, etc.: a. Continued maintenance therapy with the originally effective TKI at the same dose: The patient achieved at least stable disease (SD) or partial response (PR) during prior treatment, with progression-free survival (PFS) exceeding 6 months, and the adverse reactions were tolerable. b. Combination therapy with two TKIs: Different drugs were selected for maintenance based on distinct actionable mutations identified in the patient's tissue or peripheral blood genetic testing, OR a combination of drugs previously effective and well-tolerated was used, OR the combination therapy was chosen by referencing past tolerability.
  Arms: Physician's choice

SUMMARY:
This study is a multicenter, prospective, randomized controlled Phase II clinical trial. The primary endpoint is to evaluate the efficacy and safety of regorafenib combined with envafolimab compared to physician's choice in patients with metastatic gastrointestinal stromal tumors harboring KIT exon 17 mutations who have failed standard treatments.

DETAILED DESCRIPTION:
This multicenter, prospective, randomized, controlled phase II clinical trial aims to explore the efficacy and safety of regorafenib combined with envafolimab in treating metastatic GIST with KIT exon 17 mutation that has failed standard treatment. It also seeks to investigate the correlation between the immune microenvironment and the efficacy of immunotherapy.

The study includes patients with histologically confirmed advanced metastatic GIST containing the KIT exon 17 mutation, requiring at least one evaluable lesion. Using a block randomization method, the study is open-label and assigns patients to either the treatment group or the control group in a 1:1 ratio. The treatment group receives regorafenib combined with envafolimab, while the control group continues physician's choice until disease progression, intolerable toxicity, or voluntary withdrawal from the trial.

The governing principle for physician decision-making in the control group was selection based on prior medication tolerability, genotype, etc.:

1. Continued maintenance therapy with the originally effective TKI at the same dose: The patient achieved at least stable disease (SD) or partial response (PR) during prior treatment, with progression-free survival (PFS) exceeding 6 months, and the adverse reactions were tolerable.
2. Combination therapy with two TKIs: Different drugs were selected for maintenance based on distinct actionable mutations identified in the patient's tissue or peripheral blood genetic testing, OR a combination of drugs previously effective and well-tolerated was used, OR the combination therapy was chosen by referencing past tolerability.

A total of 100 patients are planned to be enrolled, with imaging assessments conducted at baseline and every two months during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, no gender restriction;
* Pathologically confirmed gastrointestinal stromal tumor (GIST);
* At least one measurable target lesion according to mRECIST v1.1 criteria (non-lymph node lesion with a long axis ≥ 1.0 cm or long axis ≥ 2 slide thicknesses); imaging assessment within 14 days before the first dose;
* Progression or intolerance after treatment with imatinib, sunitinib, regorafenib, or ripretinib;
* Genetic testing includes primary or secondary KIT exon 17 mutation;
* Adequate organ and bone marrow function, defined as follows:

Hematology: Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; platelet count (PLT) ≥ 75 × 10^9/L; hemoglobin (HGB) ≥ 9.0 g/dL. No use of granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), red blood cell transfusion, or platelet transfusion within 14 days before testing; Liver and kidney function: For patients without liver metastasis, total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN. For patients with liver metastasis: TBIL ≤ 1.5 × ULN; ALT and AST ≤ 5 × ULN. Kidney function: serum creatinine (Scr) ≤ 1.5 × ULN; Adequate coagulation function, defined as international normalized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 × ULN; if the patient is on anticoagulant therapy, PT should be within the intended range of the anticoagulant;

* Provide 15 paraffin-embedded tissue sections before enrollment for immune microenvironment testing;
* ECOG PS score 0-2;
* Signed informed consent.

Exclusion Criteria:

* Unable to tolerate previous regorafenib treatment or previously received immune checkpoint inhibitors;
* Pregnant or breastfeeding;
* Expected survival less than 3 months;
* Underwent major surgery or experienced significant trauma within 4 weeks before the first blood draw during the screening period, or expected to need major surgery during the study;
* Currently have active ulcers or gastrointestinal bleeding;
* History of interstitial lung disease or non-infectious pneumonia; history of active tuberculosis;
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
* Clinically diagnosed autoimmune disease; HIV or HCV positive; HBV-DNA exceeding laboratory normal range; acute CMV infection;
* Patients with central nervous system metastasis;
* Patients with other malignancies within the past five years;
* Immunosuppressed subjects, including those with known immunodeficiency; currently using systemic steroids (except for recent or current use of inhaled steroids);
* Uncontrolled hypertension: Despite aggressive antihypertensive therapy, sequential measurements show systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥100 mmHg on three consecutive occasions;
* Subjects deemed by the investigator to be unable or unwilling to comply with the study protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to disease progression or death, whichever came first, assessed up to 2 years
  Assessed by the investigator according to mRECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall Survival (OS) | Overall Survival (OS): from enrollment to death, assessed up to 2 years
  Overall Survival (OS): Assessed by the investigator according to mRECIST 1.1 criteria.
Objective Response Rate (ORR) | assessed up to 2 years
  Objective Response Rate (ORR): Assessed by the investigator according to mRECIST 1.1 criteria.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | assessed up to 2 years
  The safety parameters of this study include clinical symptoms, vital signs, physical examinations, and laboratory tests (routine, urinalysis, blood biochemistry, thyroid function, coagulation function, etc.). Adverse events (AEs) observed will be evaluated according to version 5.0 of the NCI-CTCAE, including type, incidence, severity, onset and end times, whether they are serious adverse events, and their relationship to the study drug.
  The assessment of postoperative complications includes type, incidence, and grading (based on the Clavien-Dindo classification system).

OTHER OUTCOMES:
Exploratory Study Endpoints-Correlation between the immune microenvironment of GIST and the efficacy of immunotherapy. | From enrollment to the end of the study, assessed up to 2 years
  Before enrollment, provide 15 paraffin tissue sections for the detection of immune microenvironment-related indicators, including PD-L1, CD4+ T cells, CD8+ T cells, and tumor-infiltrating lymphocytes (TILs).

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, Dr., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, 52 Fucheng Road, Beijing, Beijing Municipality, China